CLINICAL TRIAL: NCT07000565
Title: The Effect of Eye Care With Artificial Tears and Normal Saline on Ocular Surface Disease in Mechanically Ventilated Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Senanur Şimşek, Principal Investigator, Marmara University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2855458
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Ocular Surface Disease
Keywords: ocular surface disease; eye care; pediatric intensive care; nursing; artificial tears; saline
MeSH Terms: interventions — Lubricant Eye Drops; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial tears (Experimental): Every 2 hours, artificial tear solution was gently applied to the designated eye. The artificial tear product (REFRESH®) contains 5.6 mg of polyvinyl alcohol and 2.4 mg of povidone per mL and is used to maintain ocular surface moisture and reduce irritation. The eye care procedure was performed over a 5-day period while the patient remained on mechanical ventilation.
  Interventions: Other: Eye Care with Artificial Tears
- Saline (Active Comparator): Every 2 hours, saline solution (Bio-Fleks brand) was gently applied to the assigned eye for saline group.The eye care procedure was performed over a 5-day period while the patient remained on mechanical ventilation.
  Interventions: Other: Eye Care with Normal Saline

INTERVENTIONS:
Other: Eye Care with Artificial Tears — Every 2 hours, the artificial tear solution was gently applied to the designated eye for 5 days. The artificial tear product (REFRESH®) contains 5.6 mg of polyvinyl alcohol and 2.4 mg of povidone per mL and is used to maintain ocular surface moisture and reduce irritation.
  Arms: Artificial tears
Other: Eye Care with Normal Saline — Every 2 hours, the saline solution(Bio-Fleks brand) was gently applied to the designated eye for 5 days.
  Arms: Saline

SUMMARY:
The primary aim of this study is to comparatively examine the effects of eye care practices using artificial tears and normal saline on superficial ocular injuries in pediatric patients receiving mechanical ventilation in the intensive care unit. Based on the findings, the study seeks to provide evidence-based contributions to nursing practices. Additionally, it aims to identify educational strategies to enhance intensive care nurses' knowledge and practice levels and to support the development of clinical care protocols.

H0: There is no difference in the effect of eye care with normal saline and artificial tears on superficial ocular injury in mechanically ventilated pediatric patients.

H1:Eye care with normal saline is more effective than artificial tears in preventing superficial ocular injury in mechanically ventilated pediatric patients.

H2: Eye care with artificial tears is more effective than normal saline in preventing superficial ocular injury in mechanically ventilated pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 28 days to 18 years
* Receiving invasive mechanical ventilation
* Admitted to the pediatric intensive care unit
* Parent(s) or legal guardian(s) provide informed consent for participation

Exclusion Criteria:

-Having eye-related disease

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Ocular Dryness Score | Everyday for 5 days after the inclusion of participant
  Ocular dryness will be measured using the Schirmer test.The score was compared between the eye treated with artificial tears and the eye treated with normal saline.
Occurence of Ocular Surface Disease | 1 time Everyday for 5 days after the inclusion of participant
  Florescein testing will be used to evaluate the development of ocular surface disease
Change in Eyelid Closure Degree | 1 time everyday for 5 days after the inclusion of participant
  Eyelid Closure Degree was evaluated by clinical observation and scoring (e.g., staining intensity and affected area). The score was compared between the eye treated with artificial tears and the eye treated with normal saline.

CONTACTS AND LOCATIONS:
Overall Officials: Bilgi Gülseven Karabacak, MSc. PhD., Study Director — Marmara University
Locations (1):
- Istanbul University Istanbul Medical Faculty, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No